CLINICAL TRIAL: NCT05340023
Title: Proteomic Pattern Associated With the Diagnosis of Chronic Thromboembolic Pulmonary Hypertension : PROTEO-CTEPH Study.
Brief Title: Proteomic Pattern Associated With the Diagnosis of Chronic Thromboembolic Pulmonary Hypertension
Acronym: PROTEO-CTEPH
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 21CH115; ANSM (Other: 2021-A01268-33)
Record Dates: First submitted 2021-11-17; First posted 2022-04-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Pulmonary hypertension;; chronic thromboembolic pulmonary hypertension; pulmonary embolism; proteomic pattern
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Embolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample will be realized to proteomic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with suspicion of Chronic ThromboEmbolic Pulmonary Hypertension (CTEPH): * right cardiac catheterization (usual practice)
  * a blood sample (inclusion for all patients with suspicion)
  * if diagnosis of Chronic thromboembolic pulmonary hypertension confirmed a another bood sample at 6 months
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — to realize proteomic analysis.

SUMMARY:
Chronic ThromboEmbolic Pulmonary Hypertension (CTEPH) is a rare but severe complication of pulmonary embolism (PE). CTEPH is evoked in patients with persistent dyspnea. According to international guidelines, symptomatic patients with perfusion defects on lung scan and Pulmonary Hypertension (PH)-likely transthoracic echo (TTE) must be evaluated in Pulmonary Hypertension (PH)-centers with right heart catheterism, to confirm or rule out the presence of precapillary Pulmonary Hypertension (PH), and precise the group of Pulmonary Hypertension (PH).

DETAILED DESCRIPTION:
However, persistent dyspnea and perfusion defects are frequent after pulmonary embolism (PE), and the accuracy of transthoracic echo (TTE) is not great for precapillary Pulmonary Hypertension (PH).

This study proposed to seek for a specific proteomic pattern in patients admitted for a suspicion of Chronic ThromboEmbolic Pulmonary Hypertension (CTEPH).

ELIGIBILITY:
Inclusion Criteria:

* Patient with a suspicion of Chronic thromboembolic pulmonary hypertension (CTEPH) with a combination of a perfusion lung scan and transthoracic perfusion scan and transthoracic echocardiography compatible with the diagnosis (according to French recommendations)
* Patients who require a right heart catheterization.
* Patient affiliated or entitled to a social security plan
* Patient having received informed information about the study informed about the study

Exclusion Criteria:

* Patient with a normal perfusion lung scan
* Person under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to all consecutive patients admitted to the participating competence centers, provided they meet the the study, provided they meet the inclusion criteria and have no non-inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proteomic pattern associated with the diagnosis of Chronic thromboembolic pulmonary hypertension (CTEPH) | Day: 0
  Analysis of the final diagnosis retained for the patient : Chronic thromboembolic pulmonary hypertension (CTEPH) (population of interest), pre-capillary Pulmonary Hypertension (PH) other than Chronic thromboembolic pulmonary hypertension (CTEPH), post-capillary Pulmonary Hypertension (PH), no Pulmonary Hypertension (PH).

SECONDARY OUTCOMES:
Analysis of recording of hemodynamic data at diagnosis | Day: 0
  hemodynamic data : pulmonary vascular resistance, cardiac index, pulmonary arterial pressures
Analysis of recording of hemodynamic data at diagnosis | Day: 0
  hemodynamic data : pulmonary vascular resistance,
Analysis of recording of hemodynamic data at diagnosis | Day: 0
  hemodynamic data : cardiac index
Analysis of recording of hemodynamic data at diagnosis | Day: 0
  hemodynamic data : pulmonary arterial pressures
Analysis of recording of hemodynamic after 6 months of treatment | 6 months
  hemodynamic data : pulmonary vascular resistance,
Analysis of recording of hemodynamic after 6 months of treatment | 6 months
  hemodynamic data : cardiac index
Analysis of recording of hemodynamic data at diagnosis and at death | 6 months
  hemodynamic data : pulmonary arterial pressures

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BERTOLETTI, PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No